CLINICAL TRIAL: NCT05765877
Title: Neoadjuvant WX-0593 in Resectable ALK-positive or ROS1-positive Non-small Cell Lung Cancer : a Single-arm, Exploratory Trial
Brief Title: Neoadjuvant WX-0593 in Resectable ALK-positive or ROS1-positive Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pingping Song (Other)
Responsible Party: Sponsor-Investigator, Pingping Song, Department director, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WX0593-IIT-001
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer(NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- WX-0593 (Experimental): The treatment will be administrated as neoadjuvant 8 weeks before surgery. After surgical intervention the treatment will be administered up to 2 years. Treatment will be discontinued in case of unacceptable toxicity or disease progression.
  Interventions: Drug: WX-0593 Tablets

INTERVENTIONS:
Drug: WX-0593 Tablets — 60 mg of WX-0593 tablets, once daily for 7 days, followed by 180 mg of WX-0593 tablets, once daily in a 28-days cycle.

SUMMARY:
This is a single-arm, exploratory trial to evaluate the efficacy and safety of neoadjuvant WX-0593 in patients with resectable ALK-positive or ROS1- positive non-small cell lung cancer(NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer (NSCLC).
* ALK-positive or ROS1-positive NSCLC in Stage IB-IIIA (according to the 8th American Joint Committee on Cancer TNM edition), as assessed by investigator.
* Complete surgical resection of the primary NSCLC must be deemed achievable, as assessed by a MDT evaluation (which should include a thoracic surgeon, specialized in oncologic procedures).
* ECOG Performance Status of 0-1.
* At least one measurable lesion according to RECIST 1.1.
* Adequate organ and marrow function.

Exclusion Criteria:

* Prior treatment with any systemic anti-cancer therapy for NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug.
* Prior treatment with ALK TKI or ROS1 TKI.
* Prior treatment with local radiotherapy.
* Mixed small cell and NSCLC histology.
* Patients who are candidates to undergo only segmentectomies or wedge resections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Major Pathologic Response (MPR) Rate | At time of surgery
  Major pathologic response (MPR) rate is defined as percentage of residual viable tumor cells histologically detected in the resected primary tumor after surgery ≤10%.

SECONDARY OUTCOMES:
Pathologic Complete Response (pCR) Rate | At time of surgery
  Pathologic complete response (pCR) rate is defined as the percentage of participants with absence of residual tumor in lung and lymph nodes.
Resectability rate | At time of surgery
  Resectability rate is defined as the percentage of participants who were able to undergo surgery after neoadjuvant therapy.
R0 Resection rate | At time of surgery
  R0 Resection rate is defined as the percentage of participants who were able to undergo R0 Resection surgery after neoadjuvant therapy.
Objective Response Rate (ORR) | Prior to surgery
  Objective Response Rate (ORR) is defined as the percentage of participants who have a complete response (CR) or partial response (PR). Responses are according to RECIST 1.1 as assessed by investigator.
Disease Control Rate (DCR) | Prior to surgery
  Disease Control Rate (DCR) is defined as the percentage of participants who have a best overall response of CR, PR, or stable disease (SD). Responses are according to RECIST 1.1 as assessed by investigator.
Event-free survival (EFS) | 3 years postoperatively
  Event-free survival (EFS) is the length of time after initial administration the participant remains free of recurrence/progression or death, whatever the cause.
Disease-free survival (DFS) | 3 years postoperatively
  Disease-free survival (DFS) is the length of time after surgical resection the participant remains free of recurrence/progression or death, whatever the cause.
Overall Survival (OS) | 3 years postoperatively
  Overall Survival (OS) is the length of time after initial administration the participant remains alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China